CLINICAL TRIAL: NCT07057843
Title: Application Value of Sequential Nutrition Intervention Guided by Nutritional Risk Screening in CyberKnife Radiotherapy for Pancreatic Cancer
Brief Title: Sequential Nutrition Intervention for Pancreatic Cancer Patients Undergoing CyberKnife Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Feifei Wang, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023S00226
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; CyberKnife; Radiotherapy; Sequential Nutrition Intervention; Nutritional Risk Screening; Nutritional Status; Immune Function
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Study Group (Experimental): Participants received a structured, sequential nutrition intervention guided by nutritional risk screening (NRS2002). A multidisciplinary team provided the intervention, which included:
  * Pre-CyberKnife phase: Calculation of energy requirements using the Harris-Benedict formula, dietary guidance, and initiation of oral nutritional supplements (ONS). If oral intake was less than 60% of target, partial enteral (PEN) or parenteral nutrition (PPN) was administered for 7-10 days.
  * Post-CyberKnife phase: Phased re-introduction of feeding, starting with enteral nutrition via nasojejunal tube (Day 1-2) and transitioning to an oral diet (Day 3 onwards).
  * Post-discharge phase: Home energy targets were recalculated, with telephone/WeChat follow-up to ensure adherence. ONS prescribed if intake fell below 60% of targets.
  Interventions: Behavioral: Sequential Nutrition Intervention; Drug: Enteral Nutrition Emulsion
- Active Comparator: Control Group (Active Comparator): Participants received routine nutritional intervention, which consisted of dietary education focused on balanced, soft, and easily digestible meals rich in protein and other nutrients (e.g., high-protein soups).
  Interventions: Behavioral: Routine Nutritional Intervention

INTERVENTIONS:
Behavioral: Sequential Nutrition Intervention — Participants received a structured, sequential nutrition intervention guided by nutritional risk screening (NRS2002). A multidisciplinary team provided the intervention, which included:
  * Pre-CyberKnife phase: Calculation of energy requirements using the Harris-Benedict formula, dietary guidance, and initiation of oral nutritional supplements (ONS). If oral intake was less than 60% of target, partial enteral (PEN) or parenteral nutrition (PPN) was administered for 7-10 days.
  * Post-CyberKnife phase: Phased re-introduction of feeding, starting with enteral nutrition via nasojejunal tube (Day 1-2) and transitioning to an oral diet (Day 3 onwards).
  * Post-discharge phase: Home energy targets were recalculated, with telephone/WeChat follow-up to ensure adherence. ONS prescribed if intake fell below 60% of targets.
  Arms: Experimental: Study Group
Drug: Enteral Nutrition Emulsion — Fresubin (500 mL/bottle) administered at 30 mL/kg/day during the initial post-CyberKnife phase if required.
  Arms: Experimental: Study Group
Behavioral: Routine Nutritional Intervention — Participants received routine nutritional intervention, which consisted of dietary education focused on balanced, soft, and easily digestible meals rich in protein and other nutrients (e.g., high-protein soups).
  Arms: Active Comparator: Control Group

SUMMARY:
This study aims to evaluate the clinical value of a structured nutritional support program for patients with pancreatic cancer undergoing CyberKnife radiotherapy. The study compares a sequential nutrition intervention, guided by nutritional risk screening, against routine nutritional advice. The goal is to determine if the structured intervention can better improve patients' nutritional status, immune function, and quality of life, while reducing the rate of postoperative complications.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly aggressive malignancy often associated with severe malnutrition, which compromises treatment tolerance and clinical outcomes. CyberKnife radiotherapy is an effective treatment for inoperable tumors, but can still impact patient's nutritional and immune status. While nutritional support is critical, a systematic, phased approach guided by risk screening is not well-established in this patient population. This single-center, prospective, randomized controlled trial was designed to address this gap. A total of 100 patients with pancreatic cancer and malnutrition (NRS2002 score ≥3) were randomly assigned to either a study group or a control group. The control group received routine dietary education. The study group received a comprehensive sequential nutrition intervention managed by a multidisciplinary team. This intervention included initial nutritional risk screening, tailored energy and protein targets calculated using the Harris-Benedict formula, a phased protocol for nutritional support before and after CyberKnife treatment (including oral nutritional supplements, enteral, and parenteral nutrition as needed), and continued post-discharge follow-up. The hypothesis is that this structured, sequential approach will significantly improve nutritional biomarkers, enhance immune function, lead to a better quality of life, and decrease complications compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic cancer confirmed by pathological examination.
* Capacity for oral intake.
* Scheduled for CyberKnife treatment.
* Presence of malnutrition, defined by Nutritional Risk Screening 2002 (NRS2002) score ≥3.
* Expected survival >6 months.
* Karnofsky Performance Status (KPS) score ≥60.
* Provided written informed consent.

Exclusion Criteria:

* Severe cardiovascular, hepatic, or renal dysfunction.
* Concurrent malignancies of the digestive system.
* Poor treatment compliance.
* Severe ascites or edema.
* Severe cognitive impairment hindering cooperation.
* History of liver, kidney, or hematological diseases.
* Bedridden status precluding nutritional assessment.
* Long-term corticosteroid use.
* Comorbidities affecting drug metabolism or excretion (e.g., AIDS, active hepatitis).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Nutritional Indicators | Assessed at baseline (pre-intervention) and one week after intervention.
  Change from baseline in serum levels of Total Protein (TP), Transferrin (TRF), Albumin (ALB), and Prealbumin (PA).
Change in Immune Function Indicators | Assessed at baseline (pre-intervention) and one week after intervention.
  Change from baseline in peripheral blood levels of Immunoglobulin A (IgA), IgM, IgG, and T-cell subsets (CD3+, CD4+, CD8+).

SECONDARY OUTCOMES:
Change in Quality of Life (QoL) | Assessed at baseline (pre-intervention) and one week after intervention.
  Change from baseline in QoL scores, assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The score ranges from 0-100, with higher scores indicating better QoL.
Incidence of Postoperative Complications | Monitored for two weeks post-intervention.
  The number and percentage of participants experiencing postoperative complications, including malnutrition, pancreatic fistula, local pain, gastrointestinal reactions, skin burns, and hemorrhage.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China